CLINICAL TRIAL: NCT05690776
Title: Quattro® X Suture Anchor With BroadBand™ Tape Post Market Clinical Follow-up Study (Incl. Instruments)
Brief Title: PMCF Study on the Safety, Performance and Clinical Benefits Data of the Quattro X Broadband
Status: Completed | Type: Observational
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Other Study IDs: CME2021-24SM
Record Dates: First submitted 2022-12-19; First posted 2023-01-19 (Actual); Results first posted 2025-09-10 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2024-12

CONDITIONS: Rotator Cuff Tears; Rotator Cuff Injuries
Keywords: Post-Market Clinical Follow-Up Study; Medical Device; Performance; Safety; Clinical Benefits
MeSH Terms: conditions — Rotator Cuff Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients who received the Quattro X BroadBand: No specific interventions will be administered.

SUMMARY:
The study is a multicenter, retrospective and prospective, non-randomized, noncontrolled, and consecutive series post-market study. The purpose of this study is collect data confirming safety, performance and clinical benefits of the Quattro® X Suture Anchor with BroadBand™ Tape and Instruments when used in rotator cuff repair.

The primary endpoint of this study is the assessment of performance by analyzing soft tissue to bone healing in the shoulder (rotator cuff). Healing will be assessed by the investigator using PROMs and clinical outcomes of the patient. The clinical benefit will be assessed by functional outcomes measured using standard and well-established scoring systems (e.g. Constant & Murley and EQ-5D-5L) at 1 year post-operative.

The safety will be assessed by monitoring the incidence and frequency of device- and/or procedure-related adverse events.

DETAILED DESCRIPTION:
The Quattro® X Suture Anchor with BroadBand™ Tape is intended for use in rotator cuff repairs. It is intended for for the reattachment of soft tissue to bone.

Up to three sites will be involved in this study. The aim is to include a total of 109 consecutive series cases who received the Quattro® X Suture Anchor with BroadBand™ Tape. All potential study subjects will be required to participate in the Informed Consent Process.

Baseline data from the preop, intraop and immediate post-op intervals will be available in medical notes and collected retrospectively. During follow-up visits at 1 years post-op, the patient will be asked to complete patient questionnaires. Moreover, a clinical assessment will be conducted. In addition, any complications and adverse events will also be collected during these follow-up visits.

ELIGIBILITY:
Inclusion Criteria:

1. Subject treated with the Quattro® X Suture Anchor with BroadBand™ Tape for rotator cuff repair;
2. Older than 18 years and skeletally mature;
3. Willing and able to comply with the study procedures;
4. Subject is capable of understanding the doctor's explanations, following his instructions and is able to participate in the follow-up program;
5. Subject is able to read and understand the ICF and has voluntarily provided written informed consent.

Exclusion Criteria:

1. Presence of infection;
2. Insufficient or immature bone;
3. Insufficient blood supply or previous infections which may hinder the healing process;
4. Foreign body sensitivity;
5. Subject is vulnerable (prisoner, mentally incompetent or unable to understand what participation to the study entails, a known alcohol or drug abuser, anticipated to be non-compliant);
6. The subject is unwilling or unable to give consent or to comply with the follow-up program;
7. Subject meets any contraindications of the appropriate Instruction for Use.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects treated with the Quattro® X Suture Anchor with BroadBand™ Tape for rotator cuff repair, according to the IFU and who meet all of the inclusion and none of exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 106 (Actual)
Dates: Start 2022-06-17 (Actual); Primary Completion 2024-08-09 (Actual); Study Completion 2024-11-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hassan Achakri, Study Director — Zimmer Biomet
Locations (2):
- France (2):
  - Ortheo, Saint-Etienne
  - Centre Clinical, Soyaux

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Patients Who Received the Quattro X BroadBand
Started | 106
Completed | 106
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Patients Who Received the Quattro X BroadBand
Number analyzed (Participants) | 106
Age, Customized [Mean (Standard Deviation); unit: Years] — Age is recorded at the time of the surgery
  Years
    Age at surgery | 61.6 (8.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40
  Male | 66
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
BMI [Mean (Standard Deviation); unit: kg/m2] | 26.0 (3.3)
Symptom Duration [Mean (Standard Deviation); unit: days] | 349.7 (372.8)
Weight [Mean (Standard Deviation); unit: kg] | 75.2 (11.7)
Height [Mean (Standard Deviation); unit: cm] | 169.9 (8.9)
Operated Side [Count of Participants; unit: Participants]
  Left | 34
  Right | 72
Patient Employment Before Surgery [Count of Participants; unit: Participants]
  Full Time | 50
  Parti Time | 6
  Retired | 47
  Not Employed | 3
Dominant Shoulder [Count of Participants; unit: Participants]
  Left | 7
  Right | 99
Current Tobacco Use [Count of Participants; unit: Participants]
  None | 97
  Less than one pack per day | 9
Current Alcohol Use [Count of Participants; unit: Participants]
  None | 91
  Daily | 1
  Weekly | 5
  Monthly | 4
  Occasionally | 5
Constant and Murley [Mean (Standard Deviation); unit: units on a scale] — The Constant and Murley score is a 100-point functional shoulder assessment tool in which higher scores reflect increased function. The subjective variables are pain (15 points) and function (activities of daily living - sleep, work, recreation/sport; 20 points), for a total of 35 points. The objective variables are active range of motion (clinician assessment; 40 points) and strength (25 points), for a total of 65 points. The minimum score is 0 points (worst outcome), the maximum score possible is 100 points (best outcome). Population: not all patients had baseline data available
  units on a scale
    number analyzed (Participants) | 50
    (all) | 49.9 (8.4)
EQ5D [Mean (Standard Deviation); unit: units on a scale] — The EQ-5D-5L is a standardized instrument widely used to measure health status. It is a self-reported assessment about the patient's quality of life composed of two parts: a questionnaire and a visual analogue scale (VAS). The questionnaire includes 5 questions referring to mobility, self-care, daily activities, pain/discomfort and anxiety/depression. Each question can be answered in five ways, indicating no, slight, moderate, severe problems or inability to complete the task. In the derived EQ-5D-5L score, the highest score is 1 (best outcome) and the lowest score is -0.573 (worst outcome). Population: not all patients had baseline data available
  units on a scale
    number analyzed (Participants) | 50
    (all) | 0.882 (0.119)
Subjective Shoulder Value [Mean (Standard Deviation); unit: Percentage] — The Subjective Shoulder Value (SSV) is a single point, subjective estimate of a patient's condition. The patient is asked to rate the functionality of their operated shoulder on a scale of 0% - 100% of normal. Population: not all patients had baseline data available
  Percentage
    number analyzed (Participants) | 49
    (all) | 63.3 (9.1)
Prior Ipsilateral Shoulder Infection [Count of Participants; unit: Participants]
  Yes | 0
  No | 106
Prior Contralateral Shoulder Infection [Count of Participants; unit: Participants]
  Yes | 0
  No | 106
Prior Shoulder Operation(s) [Count of Participants; unit: Participants]
  Contralateral Rotator Cuff Repair | 3
  Ipsilateral Rotator Cuff Repair | 1
  No | 102
Is Contralateral Shoulder in This Study [Count of Participants; unit: Participants]
  Yes | 1
  No | 105
Functional Demand of Operated Shoulder [Count of Participants; unit: Participants]
  Low | 9
  Medium | 46
  High | 51
Concomitant Diseases [Count of Participants; unit: Participants]
  Yes | 0
  No | 106
Does The Patient Take Pain/Anti-Inflammatory Medication? [Count of Participants; unit: Participants] — Population: Not all enrolled patients had preoperative data available
  Participants
    Non-Narcotic Analgesics: number analyzed (Participants) | 49
    Non-Narcotic Analgesics: Daily | 1
    Non-Narcotic Analgesics: Weekly | 10
    Non-Narcotic Analgesics: Monthly | 2
    Non-Narcotic Analgesics: No | 36
    Narcotic Analgesics: number analyzed (Participants) | 49
    Narcotic Analgesics: Daily | 1
    Narcotic Analgesics: Weekly | 1
    Narcotic Analgesics: Monthly | 0
    Narcotic Analgesics: No | 47
    NSAIDs: number analyzed (Participants) | 49
    NSAIDs: Daily | 2
    NSAIDs: Weekly | 5
    NSAIDs: Monthly | 4
    NSAIDs: No | 38
    Steroids: number analyzed (Participants) | 49
    Steroids: Daily | 0
    Steroids: Weekly | 1
    Steroids: Monthly | 0
    Steroids: No | 48
Patient Injury [Count of Participants; unit: Participants]
  Sustained Injury | 25
  Chronic Degeneration of the Rotator Cuff | 81
Rotator Cuff Defect [Count of Participants; unit: Participants]
  Small (< 1 cm) | 7
  Medium (1-3 cm) | 63
  Large (4-5cm) | 29
  Massive (<5cm) | 7
Tendons Involved (e.g., torn) Supra; Infra [Count of Participants; unit: Participants]
  Supra, Infra | 57
  Supra, Subscap | 33
  Supra | 8
  Supra, Infra, Subscap | 7
  Subscap | 1
Procedure Performed [Count of Participants; unit: Participants]
  Single Row Repair | 1
  Double Row Repair | 105

OUTCOME MEASURES:

1. Primary Outcome: Assessment of Performance by Analyzing Soft Tissue to Bone Healing in the Shoulder (Rotator Cuff)
Description: The investigator will clinically evaluate at 1 year follow-up visit if soft tissue to bone healing has occurred by the absence of device-related revisions and re-tears that were not previously reported.
  The following question will be asked to the investigator: "Did soft tissue to bone healing occur"? If "yes" is answered, then the soft tissue to bone healing is successful, if "no" is answered, then the soft tissue to bone healing is considered unsuccessful.
Time Frame: From operation to study completion, 0-1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Patients Who Received the Quattro X BroadBand
Number analyzed (Participants) | 106
Participants
  Yes | 105
  No | 1

2. Secondary Outcome: Constant and Murley Score
Description: The Constant and Murley score is a 100-point functional shoulder assessment tool in which higher scores reflect increased function. The subjective variables are pain (15 points) and function (activities of daily living - sleep, work, recreation/sport; 20 points), for a total of 35 points. The objective variables are active range of motion (clinician assessment; 40 points) and strength (25 points), for a total of 65 points. The minimum score is 0 points (worst outcome), the maximum score possible is 100 points (best outcome).
Time Frame: From operation to study completion, 0-1 year
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Patients Who Received the Quattro X BroadBand
Number analyzed (Participants) | 106
units on a scale | 67.9 (14.7)
Statistical Analysis 1: Comparison: Patients Who Received the Quattro X BroadBand; Test type: Superiority; p < 0.0001, paired t-test; Mean Difference (Final Values) = 12.1, 95% CI 2-sided [9.2 to 15.0], Standard Deviation 10.0

3. Secondary Outcome: EQ-5D-5L Score
Description: Assessment of clinical benefits by functional outcomes measured using standard scoring systems. The EQ-5D measures 5 dimensions; mobility, self-care, usual activities, pain/discomfort, and anxiety/depression, with a total of 5 questions. It is accompanied by the patient's self-assessment with the VAS.
  Each dimension is assigned one of three discrete levels for evaluation on the day of administration:
  Level 1 - No problems, no disability Level 2 - Some problems, moderate disability Level 3 - A lot of problems, severe disability The final score is a five digit composite of the responses ranging between 33333 - 11111 with 243 possible combinations in between. In the derived EQ-5D-5L score, the highest score is 1 (best outcome) and the lowest score is -0.573 (worst outcome).
Time Frame: From operation to study completion, 0-1 year
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Patients Who Received the Quattro X BroadBand
Number analyzed (Participants) | 106
units on a scale | 0.95 (0.104)
Statistical Analysis 1: Comparison: Patients Who Received the Quattro X BroadBand; Test type: Superiority; p < 0.0001, paired t-test; Mean Difference (Final Values) = 0.09, 95% CI 2-sided [0.053 to 0.128], Standard Deviation 0.133

4. Secondary Outcome: Assessment of Safety
Description: Safety will be assessed by monitoring the incidence and frequency of device and/or procedure related adverse events
Time Frame: From operation to study completion, 0-1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Patients Who Received the Quattro X BroadBand
Number analyzed (Participants) | 106
Participants
  Patients with adverse events | 9
  Patients without adverse events | 97

5. Secondary Outcome: Subjective Shoulder Value
Description: The Subjective Shoulder Value is a patient's subjective shoulder assessment expressed as a percentage of an entirely normal shoulder.
Time Frame: From operation to study completion, 0-1 year
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | Patients Who Received the Quattro X BroadBand
Number analyzed (Participants) | 106
Percentage | 86.1 (13.3)
Statistical Analysis 1: Comparison: Patients Who Received the Quattro X BroadBand; Test type: Superiority; p < 0.0001, paired t-test; Mean Difference (Final Values) = 20.7, 95% CI 2-sided [16.9 to 24.5], Standard Deviation 13.2

6. Secondary Outcome: Pain / Anti-Inflammatory Medication
Description: Does The Patient Take Pain/Anti-Inflammatory Medication?
Time Frame: 1 year after surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Patients Who Received the Quattro X BroadBand
Number analyzed (Participants) | 106
Participants
  Non-Narcotic Analgesics: Daily | 1
  Non-Narcotic Analgesics: Weekly | 6
  Non-Narcotic Analgesics: Monthly | 1
  Non-Narcotic Analgesics: None | 98
  NSAIDs: Daily | 0
  NSAIDs: Weekly | 4
  NSAIDs: Monthly | 0
  NSAIDs: None | 102

7. Secondary Outcome: Patient Satisfaction
Description: Patient satisfaction was assessed 1 year after surgery. Possible answers were: very satisfied, satisfied, somewhat satisfied, disappointed.
Time Frame: 1 year after surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Patients Who Received the Quattro X BroadBand
Number analyzed (Participants) | 106
Participants
  Very Satisfied | 76
  Satisfied | 21
  Somewhat Satisfied | 7
  Disappointed | 2

8. Secondary Outcome: Would The Patient Have This Surgery Again?
Description: 1 year after their surgery, patients were asked if yes or no they would have the surgery again.
Time Frame: 1 year after surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Patients Who Received the Quattro X BroadBand
Number analyzed (Participants) | 106
Participants
  Yes | 85
  No | 21

ADVERSE EVENTS:
Time Frame: From surgery to last assessment 1 year postoperatively
Description: Adverse Events were collected retrospectively from the patients medical notes and prospectively at the 1 year follow up visit.
Arm/Group | Patients Who Received the Quattro X BroadBand
All-Cause Mortality (participants affected / at risk) | 0/106
Serious Adverse Events (participants affected / at risk) | 0/106
Other Adverse Events (participants affected / at risk) | 9/106
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Patients Who Received the Quattro X BroadBand (N=106)
Complex Regional Pain Syndrome (Musculoskeletal and connective tissue disorders) | 7 (7)
Re-Tear (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain and Loss of Strength (Musculoskeletal and connective tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-04-27): https://cdn.clinicaltrials.gov/large-docs/76/NCT05690776/Prot_SAP_000.pdf